CLINICAL TRIAL: NCT05037227
Title: Safety Profile Following Inactivated COVID-19 Vaccine in Healthy Adults Aged >18 Years in Indonesia
Status: Completed | Type: Observational
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Other Study IDs: COVID19-0421
Record Dates: First submitted 2021-09-06; First posted 2021-09-08 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Safety Issues

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is evaluating safety profile of COVID-19 Vaccine in healthy adults aged >18 years in Indonesia.

DETAILED DESCRIPTION:
To assess any serious systemic reaction within 30 minutes after COVID-19 vaccine immunization.

To assess systemic reaction after COVID-19 Vaccine immunization. To assess local reaction after COVID-19 Vaccine immunization. To assess any serious adverse event after COVID-19 Vaccine immunization.

ELIGIBILITY:
Inclusion Criteria:

* Clinically healthy adults aged > 18 years.
* Subjects have been informed properly regarding the study and signed the informed consent form.
* Subjects will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

* Subjects concomitantly enrolled or scheduled to be enrolled in another trial.
* Evolving mild, moderate or severe illness, especially infectious disease or fever (body temperature ≥37.5℃, measured with thermometer).
* Women who are lactating, pregnant or planning to become pregnant during the study period.
* History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection.
* Subjects who have any history of confirmed or suspected immunosuppressive or immunodeficient state, or received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products or long-term corticosteroid therapy (> 2 weeks)).
* Subjects receive any vaccination within 1 month before and after IP immunization.
* Subjects plan to move from the study area before the end of study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is involving healthy adults aged > 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Any serious adverse event occurring from inclusion until 30 minutes after the injection | Within 30 minutes after vaccination
  Number and percentage of subjects with serious systemic reactions 30 minutes after immunization.

SECONDARY OUTCOMES:
Local reaction and systemic events occurring within 30 minutes after each immunization. | Within 30 minutes after vaccination
  Number and percentage of subjects with at least one of these adverse events, solicited or not, within 30 minutes after vaccination.
Local reaction and systemic events occurring within 28 days after immunization | 28 days
  Number and percentage of subjects with at least one of these adverse events, solicited or not, within 28 days after vaccination.
Any serious adverse event during observation period. | 28 days
  Number and percentage of subjects with serious adverse event from inclusion until 28 day after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Julitasari Sundoro, MD, Principal Investigator — Indonesian Vaccine Safety Advisory Commitee
Locations (1):
- Jakarta Provincial Ministry of Health, Jakarta, DKI Jakarta, Indonesia